CLINICAL TRIAL: NCT03830216
Title: Connected Pens for Diabetes Study
Acronym: CUPID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Selective inclusion/exclusion criteria led to low enrollment which was not viable for the sponsor and site.
Sponsor: Companion Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM 2018-01
Record Dates: First submitted 2019-01-30; First posted 2019-02-05 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled treatment
Who Masked: Participant, Investigator
Masking Description: Participants in the control arm will use a blinded device. All participants will be blinded to baseline time-in-range and HbA1c measures. Investigators will be blinded to professional CGM baseline time-in-range.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): Study subjects will administer prandial insulin to manage their diabetes using a connected insulin pen and smartphone app with integrated dose calculator.
  Interventions: Device: Connected insulin pen and smartphone app
- Control Arm (Sham Comparator): Study subjects will administer prandial insulin to manage their diabetes using an inactive connected insulin pen without smartphone app.
  Interventions: Device: Inactive connected insulin pen without smartphone app

INTERVENTIONS:
Device: Connected insulin pen and smartphone app — The InPen system is a reusable pen injector for single-patient use by people with diabetes age 12 and older for the self-injection of a desired dose of insulin. The pen injector is paired with a smartphone app with dose calculator.
  Arms: Treatment Arm
Device: Inactive connected insulin pen without smartphone app — The InPen system is a reusable pen injector for single-patient use by people with diabetes age 12 and older for the self-injection of a desired dose of insulin. The pen injector is inactive and not paired with a smartphone app or dose calculator.
  Arms: Control Arm

SUMMARY:
The objective of the study is to evaluate the impact of a wireless smart insulin pen and smartphone-based bolus advisor on clinical and psychosocial outcomes in insulin-treated diabetes mellitus patients after 3 months of use.

DETAILED DESCRIPTION:
The study is a prospective, randomized, controlled treatment design. The study device will be used for multiple daily injection (MDI) therapy of insulin. The participant will interact with the study device in the uncontrolled environment of the participant's daily life. The study protocol is designed to yield meaningful data to determine clinical and psychosocial benefits of using the study device. The study will evaluate the study device as an intervention versus a control group.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is ≥ 18 years of age
2. The participant has Type 1 OR Type 2 diabetes and is being treated with intensive insulin therapy via injection for ≥ 3 months. Intensive insulin therapy is defined as at least one long acting insulin dose and two or more short acting insulin doses per day.
3. Glycated hemoglobin (HbA1c) ≥ 7.5%).
4. The participant is a current iPhone user for over 30 days.
5. Participant adjusts meal insulin doses based on carbohydrate content of meals.
6. The participant is fluent in the English language.
7. The participant and the investigator understand participant obligations and agree that the participant is willing and able to complete the study visits.
8. Patients prandial insulin need must be <30 U per meal.

Exclusion Criteria:

1. The participant has been using unblinded CGM for less than 6 months.
2. The participant uses pre-mixed insulin.
3. Current use of a smart insulin pen.
4. Use of sliding scale insulin therapy that determines insulin dosages based exclusively on specific blood glucose results
5. Used systemic oral or inhaled steroids for more than 7 days within the last 3 months
6. Oral anti-diabetic agents, with the exception of metformin
7. Injectable anti-diabetic agents other than insulin
8. The participant is legally blind or has below specified best-corrected vision level.
9. Diagnosed with any clinically significant infectious disease or major organ system disease, such as gastroparesis or renal disease (at Investigator's discretion)
10. The participant is pregnant, lactating, or plans to become pregnant in the next 6 months.
11. The participant is currently participating in another clinical study that may preclude the participant from meeting the obligations of this study.
12. The participant has any additional condition(s) (medical, social, or psychosocial) that in the investigator's opinion would warrant exclusion from the study or prevent the participant from completing or complying with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
CGM time in range | 3 months
  Percent CGM time in range (70-180 mg/dL) at 90 days, measured over 14 day period

SECONDARY OUTCOMES:
Absolute change in HbA1c | 3 months
  Average change in HbA1c from Baseline to Month 3 compared between groups
Mean sensor glucose (mg/dL) | 3 months
  Mean sensor glucose will be measured on the final blinded, professional CGM session performed at the end of the 3 month
Percent CGM time spent in hypoglycemia (70-54 mg/dl, < 54 mg/dL) | 3 months
  Percent of time spent in hypoglycemia from Baseline to Month 3 will be compared between groups
Percent CGM time spent in hyperglycemic range (>180 mg/dl, >250 mg/dL) | 3 months
  Percent of time spent in hyperglycemia from Baseline to Month 3 will be compared between groups
Change in patient reported outcomes - ADDQoL | 3 months
  The Audit of Diabetes Dependent Quality of Life (ADDQoL) Questionnaire measures diabetes-specific quality of life. The 19 items measure the impact of diabetes on specific aspects of life and the importance of these aspects of life for quality of life.
Change in patient reported outcomes - DTSQ | 3 months
  The Diabetes Treatment Satisfaction Questionnaire (DTSQ) measures diabetes treatment satisfaction. The 8 items measure treatment satisfaction and perceived frequency of hyperglycemia and hypoglycemia.
Change in patient reported outcomes - IDSS | 3 months
  The Insulin Delivery Satisfaction Survey (IDSS) measures insulin delivery device satisfaction. The 14 items measure provides a comprehensive profile of sources of device satisfaction.
Change in patient reported outcomes - HCS | 3 months
  The Hypoglycemic Confidence Scale (HCS) Hypoglycemic measures the degree to which patients feel able, secure, and comfortable regarding their ability to avoid hypoglycemia.

OTHER OUTCOMES:
Change in glycemic variability (CV and SD) | 3 months
Number of missed bolus doses and missed basal doses | 3 months
Number of SMBG measurements in participants not using CGM | 3 months
Number of insulin dose administrations | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David Ahn, MD, Principal Investigator — Hoag Memorial Hospital Presbyterian
Locations (1):
- Mary & Dick Allen Diabetes Center, Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: Undecided